CLINICAL TRIAL: NCT04669171
Title: A Global Multicenter Phase 1/2 Trial of EO2463, a Novel Microbial-Derived Peptide Therapeutic Vaccine, as Monotherapy, and in Combination With Lenalidomide and Rituximab, for Treatment of Patients With Indolent Non-Hodgkin's Lymphoma
Brief Title: A Novel Vaccine (EO2463) as Monotherapy and in Combination, for Treatment of Patients With Indolent Non-Hodgkin Lymphoma
Acronym: SIDNEY
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Enterome (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EONHL1-20
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma
Keywords: Follicular Lymphoma; Marginal Zone Lymphoma; Rituximab; Lenalidomide; Peptide-based immunotherapy
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): Safety Lead-In, Dose-Finding, Cohort, with a 3-by-3 design of EO2463 monotherapy for 6 weeks followed by addition of lenalidomide. Then, if applicable rituximab (depending on response with EO2463 + lenalidomide) will be added. Four to 18 previously treated patients with Follicular Lymphoma (FL) or Marginal Zone Lymphoma (MZL) were anticipated to be included based on safety findings.
  Interventions: Biological: EO2463; Drug: lenalidomide; Biological: rituximab
- Cohort 2 (Experimental): Anticipated approximatively 25 previously untreated patients with FL or MZL with an evaluation of EO2463 monotherapy (at the established dose in Cohort 1).
  Interventions: Biological: EO2463
- Cohort 3 (Experimental): Anticipated approximatively 6 previously untreated patients with FL or MZL with an evaluation of EO2463 (at the established dose in cohort 1) as monotherapy for 6 weeks followed by addition of rituximab if applicable (depending on response with EO2463 monotherapy).
  Interventions: Biological: EO2463; Biological: rituximab
- Cohort 4 (Experimental): Anticipated approximatively 40 patients previously treated patients with FL (or MZL). Evaluation of EO2463 (at the established dose in Cohort 1) in combination with lenalidomide from day 1 and then with addition of rituximab.
  Interventions: Biological: EO2463; Drug: lenalidomide; Biological: rituximab

INTERVENTIONS:
Biological: EO2463 — Multiple dose of EO2463
Drug: lenalidomide — D1-21 of 4-weekly cycles
  Other Names: Revlimid
  Arms: Cohort 1; Cohort 4
Biological: rituximab — Multiple doses of rituximab
  Other Names: MabThera
  Arms: Cohort 1; Cohort 3; Cohort 4

SUMMARY:
The purpose of this study is to define the recommended Phase 2 Dose, safety, tolerability, immunogenicity, and preliminary efficacy of EO2463 during monotherapy and in combination with lenalidomide and/or rituximab in patients with indolent NHL

DETAILED DESCRIPTION:
EO2463 Is an innovative cancer peptide therapeutic vaccine based on the homologies between tumor associated antigens and microbiome-derived peptides that will be administered alone and in combination with lenalidomide, rituximab, and lenalidomide/rituximab to generate safety and preliminary efficacy data in patients with indolent NHL

ELIGIBILITY:
Inclusion Criteria:

1. For inclusion in Cohorts 1 and 4 patients should have relapsed/refractory, biopsy-proven grade 1, 2 or 3A, FL or MZL, ECOG performance status 0 to 2, and have received at least one prior line of treatment. For inclusion in Cohort 4b the above applies except that patients with FL, and not patients with MZL, will be eligible for enrollment.
2. For inclusion in Cohort 2 patients should have newly diagnosed, previously untreated (radiotherapy as only prior treatment is allowed), biopsy-proven grade 1, 2 or 3A, FL or MZL. ECOG performance status 0 or 1, low tumor burden by Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria, and not be in need of standard of care therapy according to the assessment of the treating physician.
3. For inclusion in Cohort 3 patients should have newly diagnosed, previously untreated (radiotherapy as only prior treatment is allowed), biopsy-proven grade 1, 2 or 3A, FL or MZL. ECOG performance status 0 or 1, low tumor burden by GELF criteria and be in need of therapy according to the assessment of the treating physician.
4. Patients with an age ≥ 18 years old.
5. Patients who are human leukocyte antigen (HLA)-A2 positive.
6. Patients should have radiologically measurable disease with a lymph node or tumor mass greater than or equal to 1.5 cm in at least one dimension.
7. Males or non-pregnant, non-lactating, females.
8. Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other study procedures indicated in the protocol.
9. Patients having received the information sheet and who have provided written informed consent prior to any study-related procedures.

Exclusion Criteria:

1. Patients treated with dexamethasone > 2 mg/day or equivalent (i.e. 13 mg/day of prednisone, or 53 mg/day of hydrocortisone) within 14 days before the first EO2463 administration, unless required to treat an adverse event.
2. Patients with grade 3B FL or transformation to an aggressive lymphoma subtype.
3. Patients with only one prior treatment and a high-risk profile as defined by first progression of disease within 24 months of diagnosis (the exclusion is not applicable for patients with more than one prior line treatment).
4. Patients with prior exposure to EO2463.
5. Patients treated with immunotherapy (meaning immunostimulatory or immunosuppressive therapy; beside excluded, or allowed, compounds per other inclusion/exclusion criteria specifications), radionuclide therapy, radiotherapy, cytoreductive therapy, or received treatment with any other investigational agent within 28 days before the first EO2463 administration.
6. Patients to be included in Cohorts 1 and 4, and who have received rituximab or other B cell ablation therapy within 8 weeks of start of study treatment.
7. Patients to be included in Cohorts 4, who received prior CAR T-cell therapy and progressed within 6 months after this therapy.
8. Patients with abnormal laboratory values.
9. Patients with persistent Grade 3 or 4 toxicities.
10. Uncontrolled central nervous system (CNS) metastasis.
11. Other malignancy or prior malignancy with a disease-free interval of less than 3 years.
12. Patients with clinically significant disease.
13. Patients with suspected autoimmune or active autoimmune disorder or known history of an autoimmune neurologic condition (e.g. Guillain-Barré syndrome).
14. Patients with history of solid organ transplantation or allogeneic hematopoietic stem cell transplantation.
15. Pregnant and breastfeeding patients.
16. Patients with history or presence of human immunodeficiency virus and/or potentially active hepatitis B virus/hepatitis C virus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2029-05-30 (Estimated); Study Completion 2034-05-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Recommended Phase 2 Dose | Adverse Events Assessment | | Up to 24 months
  Incidences of adverse events, Treatment-Emergent Adverse events, Serious Adverse Events, Deaths, and Laboratory Abnormalities Using the National Cancer Institute-Common Terminology Criteria for Adverse events (NCI-CTCAE) V5.0.
Phase 2: Overall Response Rate | Up to 24 months
  Overall Response Rate According to the Lugano Classification 2014 during EO2463 Monotherapy
Phase 2: Complete Response Rate | Up to 24 months
  Complete remission (CR)-rate according to the Lugano Classification 2014 during therapy with the combination of EO2463/lenalidomide/rituximab.

SECONDARY OUTCOMES:
Assessment of the Immunogenicity in Relation to OMP72, OMP64, OMP65, OMP66, and UCP2 that Compose EO2463 | Up to 24 months
  Immunogenicity will be assessed by interferon-Gamma (IFN-Γ) enzyme-Linked immunospot , and/or by intracellular cytokines staining, and/or multimers staining assays.
Evaluation of Overall Survival | Up to 7 years after last patient enrolled
  The time interval from the date of first study treatment administration to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jan Fagerberg, MD, Study Director — Enterome
Locations (12):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Rochester Medical Center (URMC) - Wilmot Cancer Institute (WCI) (James P. Wilmot Cancer Center), Rochester, New York
  - University of Washington-Seattle Cancer Care Alliance, Seattle, Washington
- CHU d'Amiens-Picardie - Hopital SUD, Amiens, France
- Italy (3):
  - University of Bologna, Bologna
  - IRCCS Policlinico San Matteo Foundation - University of Pavia, Naples
  - IRCCS Policlinico San Matteo Foundation - University of Pavia, Pavia
- Spain (4):
  - University Hospital Vall d'Hebron, Institute of Oncology, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No